CLINICAL TRIAL: NCT03311555
Title: A Salvage Trial of AR Inhibition With ADT and Apalutamide With Radiation Therapy Followed by Docetaxel in Men With PSA Recurrent Prostate Cancer After Radical Prostatectomy (STARTAR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew J. Armstrong, MD (Other)
Responsible Party: Sponsor-Investigator, Andrew J. Armstrong, MD, Professor of Medicine and Surgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080868
Record Dates: First submitted 2017-09-26; First posted 2017-10-17 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Recurrent PSA-only prostate cancer following prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recurrent PSA-only non-metastatic prostate cancer (Experimental): Subjects with recurrent PSA-only prostate cancer within 4 years of prostatectomy, and a PSA of greater than 0.2 ng/mL and less than 4 ng/mL in the absence of metastatic disease on CT and bone scans.
  Interventions: Drug: Apalutamide; Drug: Androgen deprivation; Radiation: Salvage radiation therapy; Drug: Docetaxel

INTERVENTIONS:
Drug: Apalutamide — 240mg tablet daily for 36 weeks
  Other Names: ARN-509; JNJ-56021927
Drug: Androgen deprivation — ADT will consist of treatment with a GnRH agonist or antagonist per physician and institutional preference. Either leuprolide acetate (Lupron Depot, 22.5 mg or 45 mg IM), triptorelin pamoate (Trelstar, 11.25 mg or 22.5 mg IM), goserelin acetate (Zoladex, 10.8mg SC) or degarelix (Firmagon 120 mg or 240 mg SC) will be administered monthly, every 3 months, or every 6 months, depending on institutional standards, for 36 weeks total.
Radiation: Salvage radiation therapy — On week 9 (+/- 28 days), subjects will begin salvage radiation therapy to the prostate bed. The total dose to the prostate bed must be 66-74 Gy in 1.8-2 Gy daily fractions over a total of 6-8 weeks
Drug: Docetaxel — About 4 weeks (+/- 2 weeks, pending recovery of adverse events from radiation to Grade 2 or less) after completing radiation, patients will start docetaxel 75mg/m2 intravenously, every 3 weeks for 6 cycles.

SUMMARY:
The purpose of this study is to describe the rate of 3-year progression free survival in men with recurrent PSA-only disease after prostatectomy, who receive combined apalutamide (ARN-509) and standard ADT with salvage radiation therapy followed by docetaxel, ADT, and apalutamide, AND who have had testosterone recovery to >100 ng/dl at 36 months. The hypothesis is that AR inhibition with apalutamide added to standard salvage external beam radiation with androgen deprivation therapy, as well as the addition of 6 cycles of docetaxel, will further prolong progression free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed diagnosis of prostate adenocarcinoma. Variants of prostate cancer, including neuroendocrine features and small cell carcinoma of the prostate, are not permitted.
2. Gleason sum of 7 (with pT3 disease or positive margins or positive nodes [4 or fewer]), 8, 9, or 10 based on the radical prostatectomy specimen
3. PSA relapse within 4 years of prostatectomy defined by persistently detectable or rising PSA after surgery.
4. Evidence of disease recurrence or progression as evidenced by a PSA > 0.20. This requires 2 consecutive rises in PSA, at least 1 week apart, over the post-prostatectomy nadir OR one PSA value above 0.20 ng/mL IF the patient failed to achieve a post-prostatectomy nadir of < 0.2 ng/mL.
5. Age ≥ 18 years
6. Karnofsky performance status ≥ 80
7. Adequate laboratory parameters

   * Adequate bone marrow function: ANC ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hb >9g/dL
   * AST/SGOT and ALT/SGPT ≤ 2.5 x Institutional Upper Limit of Normal (ULN)
   * Serum bilirubin ≤ 1.5 x Institutional ULN (In subjects with Gilbert's syndrome, if total bilirubin is > 1.5xULN, measure direct and indirect bilirubin and patient is eligible if direct bilirubin ≤ 1.5xULN).
   * Glomerular filtration rate (either estimated or calculated from 24-hour urine collection) ≥ 45 mL/min
   * Serum potassium ≥3.5 mmol/L
8. A minimum of 4 weeks from any major surgery prior to Cycle 1 Day 1.
9. Ability to swallow, retain, and absorb oral medication.
10. Ability to understand and the willingness to sign a written informed consent document.
11. Must use a condom if having sex with a pregnant woman.
12. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration.

Exclusion Criteria:

1. Radiographic evidence of metastatic disease. Patients with node-positive disease (≤4 positive nodes) at the time of radical prostatectomy are eligible. Patients with pelvic nodes less than 1.5 cm by short axis at the time of screening are eligible. Patients with any enlarged lymph nodes in the retroperitoneum or above the aortic bifurcation or with pelvic nodes ≥ 1.5 cm must be excluded.
2. PSA ≥ 4.0 ng/mL.
3. Testosterone level ≤ 100 ng/dL.
4. More than 1 month of prior hormone exposure or hormone exposure within 30 days of enrollment (up to 1 month of prior LHRH agonist and/or anti-androgen therapy as neoadjuvant therapy prior to prostatectomy is allowed). Prior enzalutamide, apalutamide, ketoconazole, abiraterone, or TAK700 for prostate cancer are prohibited. Prior antiandrogen therapy (including but not limited to bicalutamide, flutamide, nilutamide, enzalutamide, and apalutamide) and prior estrogen therapy (including estrogen patch) are not allowed. All investigational agents are prohibited within 30 days of enrollment.
5. The following medications are prohibited within 2 weeks of enrollment and while on study drug:

   * 5 α-reductase inhibitors (finasteride, dutasteride);
   * Biologic or other agents with anti-tumor activity against prostate cancer;
   * Systemic glucocorticoids greater than the equivalent of 10 mg per day of prednisone; oPremedication with systemic glucocorticoids greater than the equivalent of 10 mg per day of prednisone is permitted prior to docetaxel infusions.
   * Androgens (testosterone, dihydroepiandrosterone [DHEA], etc.)
6. Prior immunotherapy including sipuleucel-T.
7. Prior systemic chemotherapy (docetaxel, cabazitaxel, estramustine, other cytotoxic agents)
8. History of solid organ or stem cell transplantation.
9. History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, prior head or traumatic brain injury with loss of consciousness, prior or current space-occupying lesion in the brain). Also, history of loss of consciousness or transient ischemic attack within 12 months of Day 1 visit.
10. Known or suspected brain metastasis or active leptomeningeal disease.
11. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.
12. Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to enrollment
13. Sustained uncontrolled hypertension (>150/90 average over 1 week) despite optimal medical management
14. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of apalutamide or increase the risk of radiation (e.g., uncontrolled nausea, vomiting, diarrhea, malabsorption syndromes, prior small bowel resection, or inflammatory bowel disease).
15. Patients who have received prior prostate or pelvic radiotherapy, including external beam or brachytherapy.
16. Patients who have not recovered from side effects of prior systemic therapy prior to Cycle 1 Day 1.
17. Use of medications known to lower the seizure threshold within 4 weeks prior to study entry.
18. Patients unable or unwilling to abide by the study protocol or cooperate fully with the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tian Zhang, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - GU Research Network / Urology Cancer Center, Omaha, Nebraska
  - Weill Cornell Medical Center, New York, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Univesity, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Started | 39
Completed | 38
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 34
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at 36 Months (3 Years)
Description: The percentage of subjects with testosterone >100 ng/dl at 36 months post-Cycle 1 Day 1 without one or more of the following: Serum PSA value of 0.2 ng/mL or more above the post-radiotherapy PSA nadir and confirmed (at least) 4 weeks later by a second PSA measurement higher than the first by any amount; Continued rise in the PSA level following study treatment if no nadir is experienced, defined as 2 rising values greater than the baseline PSA and separated by at least 4 weeks; Evidence of clinical progression or initiation of systemic therapy for progressive disease; Death
Time Frame: up to 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
percentage of participants | 69.2 [56.5 to 86.5]

2. Secondary Outcome: Number of Participants With a PSA of <0.1 ng/mL and Testosterone Recovery at 12 Months Post-Cycle 1 Day 1
Description: Testosterone recovery defined as testosterone >100 ng/dl
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
Participants | 38

3. Secondary Outcome: Percentage of Participants With a PSA of <0.1 ng/mL and Testosterone Recovery at 24 Months Post-Cycle 1 Day 1
Description: Testosterone recovery defined as testosterone >100 ng/dl
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
percentage of participants | 67

4. Secondary Outcome: Percentage of Participants With a PSA of <0.1 ng/mL and Testosterone Recovery at 36 Months Post-Cycle 1 Day 1
Description: Testosterone recovery defined as testosterone >100 ng/dl
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
percentage of participants | 69

5. Secondary Outcome: Biochemical Progression-free Survival (PFS) at 36 Months (3 Years)
Description: Percentage of participants still alive without disease progression based on PSA (prostate-specific antigen) only. Must have serum PSA value of 0.2 ng/mL or more above the post-radiotherapy PSA nadir and confirmed (at least) 4 weeks later by a second PSA measurement higher than the first by any amount.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
percentage of participants | 69.2 [56.5 to 86.5]

6. Secondary Outcome: Median PSA Nadir Value
Description: Median PSA nadir value
Time Frame: 36 months
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
ng/mL | NA (NA) — Below the level of detection.

7. Secondary Outcome: Time to Testosterone Recovery
Description: Testosterone recovery defined as testosterone >100 ng/dl
Time Frame: up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
months | 15 [13 to 17]

8. Secondary Outcome: Percentage of Participants With Adverse Events as Assessed by CTCAE v4.0
Description: To describe the safety, feasibility and tolerability profile of combination apalutamide, ADT, and radiation therapy followed by apalutamide, ADT, and docetaxel as assessed by NCI common toxicity scales
Time Frame: up to 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
percentage of participants | 100

9. Secondary Outcome: Percentage of Participants Completing All Treatments
Description: To describe the percentage of participants completing all treatments including salvage radiation therapy and 6 cycles of docetaxel
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
Number analyzed (Participants) | 39
percentage of participants | 97.4

ADVERSE EVENTS:
Time Frame: 36 months
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov
Arm/Group | Recurrent PSA-only Non-metastatic Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 4/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recurrent PSA-only Non-metastatic Prostate Cancer (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Hematoma (Vascular disorders) | 1
Pelvic infection (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recurrent PSA-only Non-metastatic Prostate Cancer (N=39)
Injury, poisoning and procedural complications - Other, Specify (Injury, poisoning and procedural complications) | 1
Anemia (Blood and lymphatic system disorders) | 25
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, Specify (Ear and labyrinth disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 3
Dry eye (Eye disorders) | 1
Eye disorders - Other, Specify (Eye disorders) | 3
Photophobia (Eye disorders) | 1
Watering eyes (Eye disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 2
Anal pain (Gastrointestinal disorders) | 3
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 17
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, Specify (Gastrointestinal disorders) | 6
Hemorrhoids (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 17
Oral dysesthesia (Gastrointestinal disorders) | 3
Proctitis (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 3
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Edema face (General disorders) | 1
Edema limbs (General disorders) | 12
Fatigue (General disorders) | 35
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 6
General disorders and administration site conditions - Other, Specify (General disorders) | 8
Infusion related reaction (General disorders) | 5
Localized edema (General disorders) | 2
Malaise (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 7
Allergic reaction (Immune system disorders) | 1
Infections and infestations - Other, Specify (Immune system disorders) | 1
Mucosal infection (Immune system disorders) | 2
Otitis externa (Immune system disorders) | 1
Papulopustular rash (Immune system disorders) | 2
Pelvic infection (Immune system disorders) | 1
Penile infection (Immune system disorders) | 1
Skin infection (Immune system disorders) | 4
Upper respiratory infection (Immune system disorders) | 2
Urinary tract infection (Immune system disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 32
Platelet count decreased (Investigations) | 7
Weight gain (Investigations) | 6
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 33
Alkalosis (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Musculoskeletal and connective tissue disorders) | 9
Hypercalcemia (Musculoskeletal and connective tissue disorders) | 1
Hypoalbuminemia (Musculoskeletal and connective tissue disorders) | 2
Hypokalemia (Musculoskeletal and connective tissue disorders) | 12
Hypomagnesemia (Musculoskeletal and connective tissue disorders) | 1
Hyponatremia (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other Specify (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 2
Concentration impairment (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 6
Dysesthesia (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 23
Headache (Nervous system disorders) | 9
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 4
Nervous system disorders - Other, Specify (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 14
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5
Presyncope (Nervous system disorders) | 1
Radiculitis (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 8
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 18
Libido decreased (Psychiatric disorders) | 3
Psychiatric disorders - Other, Specify (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Renal and urinary disorders - Other, Specify (Renal and urinary disorders) | 4
Urinary frequency (Renal and urinary disorders) | 18
Urinary incontinence (Renal and urinary disorders) | 9
Urinary retention (Renal and urinary disorders) | 3
Urinary tract pain (Renal and urinary disorders) | 9
Urinary urgency (Renal and urinary disorders) | 15
Breast pain (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 2
Perineal pain (Reproductive system and breast disorders) | 1
Testicular disorder (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 30
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 10
Nail discoloration (Skin and subcutaneous tissue disorders) | 6
Nail loss (Skin and subcutaneous tissue disorders) | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 13
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 13
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other, Specify (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 39
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3
Phlebitis (Vascular disorders) | 2
Superficial thrombophlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT03311555/Prot_SAP_000.pdf